CLINICAL TRIAL: NCT02090088
Title: Nplate® Pregnancy Exposure Registry (NPER)
Brief Title: Nplate® Pregnancy Exposure Registry
Acronym: NPER
Status: Terminated | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20080046
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Birth Defect; Spontaneous Abortions; Low Birth Weight
MeSH Terms: conditions — Congenital Abnormalities; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All Subjects: All Subjects
  Interventions: Drug: Not applicable- observational study

INTERVENTIONS:
Drug: Not applicable- observational study

SUMMARY:
US study to estimate the prevalence at birth of major birth defects (ie, those that cause significant functional or cosmetic impairment, require surgery, or are life-limiting) in children born to mothers who have received Nplate® therapy at any time during the pregnancy.

DETAILED DESCRIPTION:
The purpose of the NPER is to monitor pregnancies exposed to Nplate® and to detect and record serious adverse events in infants up to one year after birth. The lack of adequate human fetal safety data for Nplate® makes the NPER an important component of the pharmacovigilance program on the safety of this drug. With respect to fetal outcome, it is important to evaluate the spectrum of outcomes that may be relevant to a medication exposure during pregnancy, and these include both easily recognizable defects that are visible at birth, as well as more subtle or delayed defects that may not be readily identifiable without special expertise and observation beyond the newborn period.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be currently pregnant women residing in the US who: Have had any exposure to Nplate® at any time during the pregnancy, which is defined as the period between first day of the last menstrual period (LMP) (ie, within two weeks of conception) up to any date before the date of delivery or end of the pregnancy. The date of conception will be defined as fourteen days prior to the next expected menstrual period for women who report a regular menstrual cycle. If the date of the first day of the LMP is unclear, or if the estimated date of conception as determined by a first-trimester ultrasound differs by more than one week from the date as determined by the first day of LMP, the first-trimester ultrasound-derived date will be used to estimate the timing of exposure to Nplate®, as well as timing of enrollment. If neither a clear date of the first day of the LMP nor a first-trimester ultrasound is available, the estimated date of conception for purposes of enrollment will be determined by best estimate of the woman's prenatal care provider.
* Agree to enroll at any time from the estimated date of conception up to any date before the date of delivery or end of the pregnancy and who have not already had prenatal diagnosis of any major structural birth defect in the current pregnancy prior to enrollment.
* Agree to provide consent for participation in the registry including follow-up interviews.

Exclusion Criteria:

* Subjects will be ineligible for study participation if any of the following apply:
* Exposure to Nplate® did not occur during pregnancy.
* Prior knowledge of prenatal diagnosis of a birth defect. Patients who fall under this category will be encouraged to call the Amgen PSP toll free number for enrollment and follow-up.
* Cases reported to the NPER after completion of the exposed pregnancy. Patients who fall under this category will be encouraged to call the Amgen PSP toll free number for enrollment and follow-up.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of two cohorts of women and their offspring who reside in the U.S. The exposed cohort is defined as pregnant women who have received at least one dose of Nplate® during pregnancy and their offspring up to one year of age. The unexposed cohort is defined as women unexposed to Nplate® during pregnancy matched on disease status (cITP) and age (childbearing) to the exposed. In order to provide context for any possible Nplate® exposed women without cITP, comparators from published literature will be used.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The registry was initiated in May 2009. The first participant enrolled in June 2010 and the last participant enrolled in December 2013.
  Eligible participants were currently pregnant women residing in the United States who had any exposure to Nplate at any time during pregnancy.
Pre-assignment Details: The Nplate® Pregnancy Exposure Registry (NPER) was to continue the follow-up of enrollees until April 2016; however, the NPER was terminated on 24 January 2014 because of the low number of participants enrolled.
Groups:
- All Participants: Pregnant woman who had any exposure to Nplate® at any time during pregnancy.
Period: Overall Study
Arm/Group | All Participants
Started | 4
Gave Birth | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Born With Major Birth Defects
Description: An external, independent Congenital Malformation Adjudication Panel (CMAP) comprised of two clinical dysmorphologists and/or teratologists organized malformations based upon organ system and embryology, and determined whether structural defects were major or minor according to a modification of the Metropolitan Atlanta Congenital Defects Program (MACDP) birth defect classification system. A major structural defect is defined as a defect which has either cosmetic or functional significance to the child (eg, a cleft lip), require surgery, or are life-limiting).
Time Frame: At birth
Population: Children born to enrolled participants during the study
Measure: Number; unit: children
Arm/Group | All Participants
Number analyzed (Participants) | 4
children | 0

2. Secondary Outcome: Number of Children Born With Any 3 or More Minor Birth Defects
Description: An external, independent Congenital Malformation Adjudication Panel (CMAP) comprised of two clinical dysmorphologists and/or teratologists organized malformations based upon organ system and embryology, and determined whether structural defects were major or minor according to a modification of the Metropolitan Atlanta Congenital Defects Program (MACDP) birth defect classification system. A minor structural defect is defined as a defect which occurs in less than 4% of the population but which has neither cosmetic nor functional significance to the child (eg, complete 2,3 syndactyly of the toes).
Time Frame: At birth
Population: Children born to enrolled participants during the study
Measure: Number; unit: children
Arm/Group | All Participants
Number analyzed (Participants) | 4
children | 0

3. Secondary Outcome: Number of Children Born With a Specific Pattern of Minor Birth Defects
Description: Only those infants who have received medical evaluation and who have three or more minor defects will be considered "affected" for purposes of the evaluation of a pattern of minor defects.
Time Frame: At birth
Population: Children born with 3 or more minor birth defects
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Spontaneous and Elective Abortions or Stillbirths
Description: Number of each of spontaneous abortions, elective abortions, and stillbirths among mothers who received Nplate® therapy at any time during the pregnancy.
Time Frame: 9 months (during pregnancy)
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 4
participants
  Spontaneous abortions | 0
  Elective abortions | 0
  Stillbirths | 0

5. Secondary Outcome: Number of Children With Preterm Birth or Low Birth Weight
Description: Number of children with preterm birth (<37 weeks gestation) or low birth weight (<2,500 grams) among children born to mothers who have received Nplate® therapy at any time during the pregnancy.
Time Frame: At birth
Population: Children born to enrolled participants during the study
Measure: Number; unit: children
Arm/Group | All Participants
Number analyzed (Participants) | 4
children
  Preterm birth | 1
  Low birth weight | 1

6. Secondary Outcome: Number of Children Born With Intrauterine Growth Restriction
Description: Number of children born with intrauterine growth restriction (weight, length or head circumference less than tenth percentile for sex and gestational age) among mothers who have received Nplate® therapy at any time during the pregnancy.
Time Frame: At birth
Population: Children born to enrolled participants during the study
Measure: Number; unit: children
Arm/Group | All Participants
Number analyzed (Participants) | 4
children | 1

7. Secondary Outcome: Number of Infants With Adverse Events
Description: In the first year of life, the incidence of all serious adverse events, as well as of nevi (birthmarks) and angiomata (benign tumors with blood vessels or lymph vessels), among infants whose mothers received Nplate® therapy at any time during the pregnancy.
Time Frame: 12 months from birth
Population: Children born to enrolled participants during the study
Measure: Number; unit: infants
Arm/Group | All Participants
Number analyzed (Participants) | 4
infants
  Serious adverse events | 2
  Nevi | 0
  Angiomata | 0

8. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Throughout pregnancy and for up to 6 weeks after delivery
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 4
participants | 4

ADVERSE EVENTS:
Time Frame: Women were assessed during pregnancy (up to 9 months) and up to 6 weeks after delivery; Infants were assessed for up to 1 year after birth.
Groups:
- Infants: Infants who were born to enrolled participants during the study.
Arm/Group | All Participants | Infants
Serious Adverse Events (participants affected / at risk) | 4/4 | 2/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=4) | Infants (N=4)
Caesarean section (Surgical and medical procedures) | 1 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 2 | 1
Therapeutic response decreased (General disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Placental Infarction (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature Delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Intraventricular Haemorrhage (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The number of infants born to participants was too low to draw conclusions or make comparisons to the Systematic Tracking of Real Kids (STORK) analysis or to the background rates of congenital anomalies or preterm infants in the general population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.